CLINICAL TRIAL: NCT00003441
Title: Phase II Study of MGI-114 (NSC# 683863) Administered Intravenously for Five Days Every 28 Days to Patients With Metastatic Colorectal Cancer
Brief Title: Irofulven in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM97-308; P30CA016672 (NIH); U01CA070172 (NIH); MDA-DM-97308 (Other: UT MD Anderson Cancer Center); NCI-T97-0113; CDR0000066469 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; 6-hydroxymethylacylfulvene; MGI-114; Irofulven
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irofulven (Experimental): 6-hydroxymethylacylfulvene (MGI-114) IV over 5 minutes daily for 5 consecutive days every 28 day cycle.
  Interventions: Drug: Irofulven (MGI-114)

INTERVENTIONS:
Drug: Irofulven (MGI-114) — IV over 5 minutes daily for 5 consecutive days. Courses repeated every 28 days. Minimum treatment period is 2 courses.
  Other Names: 6-hydroxymethylacylfulvene; MGI-114

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of 6-hydroxymethylacylfulvene (MGI-114) when given daily for 5 days every 28 days to patients with metastatic adenocarcinoma of the colon or rectum. II. Evaluate the qualitative and quantitative toxicities of MGI-114 given on this schedule in this patient population.

OUTLINE: Patients receive 6-hydroxymethylacylfulvene (MGI-114) IV over 5 minutes daily for 5 consecutive days. Courses are repeated every 28 days. The minimum treatment period is 2 courses. Treatment continues indefinitely in the absence of unacceptable toxic effects or disease progression. Patients are followed at the end of every other course while on the study, and then every 3 months thereafter until death.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study within 6-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic adenocarcinoma of the colon or rectum Bidimensionally measurable lesions Sentinel lesions outside the field of any prior radiation therapy No confirmed or suspected brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-1 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No active congestive heart failure No uncontrolled angina At least 6 months since prior myocardial infarction No uncontrolled hypertension Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent serious infection No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix No overt psychosis or mental disability No life threatening illness (unrelated to tumor)

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiation therapy and recovered No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: At least 28 days since prior administration of any investigational drug No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 1998-08; Primary Completion 2000-11-08 (Actual); Study Completion 2000-11-08 (Actual)

PRIMARY OUTCOMES:
Antitumor Activity of MGI-114 | Every 28 day cycle

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Hoff, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org